CLINICAL TRIAL: NCT04473989
Title: The Effect of Weekly Injection of Teriparatide on the Healing of Distal Radius Fracture in a Double-blind, Randomized Controlled Clinical Trial
Brief Title: Weekly Use of Teriparatide to Accelerate Healing of Distal Radius Fracture
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M2020207
Record Dates: First submitted 2020-07-12; First posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-06

CONDITIONS: Colles' Fracture
MeSH Terms: conditions — Colles' Fracture | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Injection product without active teriparatide
  Interventions: Drug: Placebo
- PTH 40ug/w (Experimental): Injection product with active teriparatide
  Interventions: Drug: recombinant teriparatide for injection

INTERVENTIONS:
Drug: recombinant teriparatide for injection — weekly subcutaneous administration of 40 ug
  Other Names: Xinfutai
  Arms: PTH 40ug/w
Drug: Placebo — weekly subcutaneous administration of 40 ug
  Other Names: Xinfutai placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effect of weekly dosing strategy on fracture healing.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women aged 45-75 (at least 2 years after menopause)
2. With primary osteoporosis
3. Patients with Colles fractures with a fracture time of no more than 7 days
4. conservative treatment after fracture (closed reduction and immobilization)
5. no multiple fractures
6. Informed well and agree to participate in this clinical trial

Exclusion Criteria:

1. Combine other physical diseases, including diabetes, severe hypertension, autoimmune diseases, heart, liver and kidney diseases, malignant tumors, mental illnesses, and other diseases that doctors believe may affect the healing process.
2. In addition to primary osteoporosis, any disease affecting bone metabolism or treatment response, including serum PTH>65pg/ml, 25-hydroxyvitamin D<20ng/ml, alkaline phosphatase>135U/L, history of bone tumor, Paget disease, history of radiotherapy
3. The fracture site has a history of trauma or surgery, affecting the function of the wrist or forearm
4. Those who are allergic to PTH or any excipients
5. Currently receiving anti-osteoporosis treatment or receiving other anti-osteoporosis treatment during the trial
6. Contraindication of teriparatide including hyperparathyroidism, severe renal insufficiency, hypercalcemia, etc.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women
Enrollment: 80 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
The median time of radiographic healing | 0-14 weeks
  A score of 13 by Modified Radiographic Union Scale for Tibia fractures (mRUST) scoring system would provide a confident assessment of union

SECONDARY OUTCOMES:
Patient-Rated Wrist Evaluation | 0, 4, 6, 8, 10, 12, 14 and 16 weeks
  A 15-item questionnaire(PRWE) that rates wrist-related pain and disability in functional activities. The scores range from 0 (no disability) to 100 (severest disability).
Grip strength | 6, 8, 10, 12, 14, and 16 weeks
  Grip strength will be assessed by a dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Chunli Song, M.D.; Ph. D., Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aspenberg P, Genant HK, Johansson T, Nino AJ, See K, Krohn K, Garcia-Hernandez PA, Recknor CP, Einhorn TA, Dalsky GP, Mitlak BH, Fierlinger A, Lakshmanan MC. Teriparatide for acceleration of fracture repair in humans: a prospective, randomized, double-blind study of 102 postmenopausal women with distal radial fractures. J Bone Miner Res. 2010 Feb;25(2):404-14. doi: 10.1359/jbmr.090731. PMID 19594305
- [Background] Ebata S, Takahashi J, Hasegawa T, Mukaiyama K, Isogai Y, Ohba T, Shibata Y, Ojima T, Yamagata Z, Matsuyama Y, Haro H. Role of Weekly Teriparatide Administration in Osseous Union Enhancement within Six Months After Posterior or Transforaminal Lumbar Interbody Fusion for Osteoporosis-Associated Lumbar Degenerative Disorders: A Multicenter, Prospective Randomized Study. J Bone Joint Surg Am. 2017 Mar 1;99(5):365-372. doi: 10.2106/JBJS.16.00230. PMID 28244906
- [Background] Zhang W, Zhu J, Ma T, Liu C, Hai B, Du G, Wang H, Li N, Leng H, Xu Y, Song C. Comparison of the effects of once-weekly and once-daily rhPTH (1-34) injections on promoting fracture healing in rodents. J Orthop Res. 2018 Apr;36(4):1145-1152. doi: 10.1002/jor.23750. Epub 2017 Nov 20. PMID 28960481
- [Derived] Zhu J, Zhang C, Jia J, Yuan W, Zhang M, Leng H, Song C. Effect of weekly teriparatide injections on osteoporotic fracture healing: protocol for a double-blind, randomised controlled trial. BMJ Open. 2021 Apr 1;11(4):e043137. doi: 10.1136/bmjopen-2020-043137. PMID 33795297